CLINICAL TRIAL: NCT06076941
Title: Effects of Education on Oral and Dental Health Behaviors and Knowledge Levels of Pregnant Women
Brief Title: Effect Of Oral And Dental Health Education In Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Seda Guray, Research Assistant, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: TarsusU2
Record Dates: First submitted 2023-09-24; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Pregnancy
Keywords: Prengnancy; oral and dental health; Education; knowledge and behavior
MeSH Terms: conditions — Behavior | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The study was conducted as a randomized controlled experimental study to determine the effect of the education given to pregnant women on their oral and dental health behaviors and knowledge levels. With the power analysis, α = 0.05, β = 0.20, 1-β = 0.80, a total of 60 pregnant women, 30 in the experimental group and 30 in the control group were included (the power of the test was found as p = 0.8056).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Experimental): Pregnant women in the experimental group were given oral and dental health education in groups of maximum five, and the forms were filled out before and one month after the education.
  Interventions: Other: Education
- Control (No Intervention): No intervention was made to the pregnant women in the control group, and the forms were completed before and one month after the training.

INTERVENTIONS:
Other: Education — Before the training was given to the pregnant women in the experimental group who agreed to participate in the study, the Introductory Information Form, the Form for Assessing Pregnant Women's Behaviors Towards Oral and Dental Health, and the Form for Assessing Pregnant Women's Knowledge Levels Towards Oral and Dental Health were applied by face-to-face interview method. The application of the forms took 20-30 minutes. Then, a training time was planned on a suitable date for the pregnant women.
  In order to ensure the effectiveness of the training, to answer the questions of the pregnant women effectively and to be able to direct them to the dentist in line with their needs, the training was applied in groups of maximum five people. Lecture, question and answer and demonstration methods were used in the training.
  One month after the training, the necessary forms were applied to the pregnant women and the study was terminated.
  Arms: Education

SUMMARY:
The study was conducted as a randomized controlled experimental study to determine the effect of the education given to pregnant women on their oral and dental health behaviors and knowledge levels.

DETAILED DESCRIPTION:
In line with these results, it is recommended that midwives should determine the behaviors and knowledge levels of pregnant women regarding oral and dental health within the scope of primary health care services, provide trainings to increase their knowledge and awareness on the subject, refer them to treatment in the presence of problems, and expand these services within the health system.

ELIGIBILITY:
Inclusion Criteria:

* Being in the first trimester of pregnancy
* Being 19-44 years old,
* Being able to read and write turkish,
* Being a healthy pregnant woman who agrees to participate in the study

Exclusion Criteria:

* Having a risky pregnancy,
* Can't speak or understand Turkish
* Women with intellectual disability
* Serious mental disorders will be excluded from the study.

Ages: 19 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Form for Assessment of Knowledge Levels of Pregnant Women Regarding Oral and Dental Health | up to 24 weeks
  This form was developed by the researcher by reviewing the literature to determine the knowledge levels of pregnant women about oral and dental health and their educational needs in this direction. The form includes 22 questions assessing the importance of dietary habits for oral and dental health, visiting a dentist during pregnancy, dental and gum treatment during pregnancy, and dental x-rays during pregnancy. The form is evaluated by giving "1 point" for correct answers and "0 point" for incorrect answers in line with the answer key specified in Appendix 4. The lowest score that can be obtained from the form is 0 and the highest score is 22. High scores indicate a high level of knowledge.
Form for Assessment of Oral and Dental Health Behaviors of Pregnant Women | up to 24 weeks
  This form was developed by the researcher by reviewing the literature to determine the oral and dental health behaviors of pregnant women. The form consists of 16 questions evaluating the behaviors of pregnant women such as current dental health status, frequency of tooth brushing, tooth brushing technique, fluoride toothpaste use, frequency of flossing and frequency of toothbrush replacement.
Pregnant Women's Education Satisfaction Evaluation Form | up to 24 weeks
  This form was prepared by the researcher to evaluate the effectiveness and benefits of the training and the opinions of the pregnant women in the experimental group after the training.
Descriptive Information Form | up to 24 weeks
  This form was developed by the researcher and consisted of two parts: sociodemographic characteristics and obstetric characteristics of pregnant women. Sociodemographic characteristics included questions such as age, education level, employment status, spouse's employment status, income level and family type. Obstetric characteristics included information on the number of pregnancies, number of living children and gestational week. There are 14 questions in the descriptive information form

CONTACTS AND LOCATIONS:
Overall Officials: Özlem DURAN AKSOY, Study Director — Cumhuriyet University
Locations (1):
- Tarsus University, Tarsus, Takbaş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No